CLINICAL TRIAL: NCT06757153
Title: Clinical Study on the Safety and Efficacy of NRG-103 Injection in the Treatment of Recurrent Glioblastoma Patients
Brief Title: Safety and Efficacy of NRG-103 Injection in the Treatment of Recurrent Glioblastoma Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhiqiang Li, Principal Investigator, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRG103001; ChiCTR2400093705 (Other Grant/Funding Number: NEURAGEN, Suzhou, China)
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma (GBM)
Keywords: Glioblastoma;Oncolytic virus;NRG103;Trans-differentiation;
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NRG-103 (Experimental): NRG-103 is an innovative gene therapy drug developed based on the in situ trans-differentiation technology. Through multiple mutation modifications of the adenovirus genome, it can enhance the specific recognition and killing effect of oncolytic virus on GBM tumor cells without being limited by tumor gene phenotype, and regulate the immune microenvironment to induce stronger anti-tumor immune response. In addition, the two transcription factors expressed on NRG-103 can efficiently transdifferentiate residual GBM tumor cells into non tumor like neuronal cells, in order to achieve the goal of delaying tumor recurrence and long-term survival.
  Interventions: Drug: NRG-103

INTERVENTIONS:
Drug: NRG-103 — NRG-103 is an oncolytic virus, which can kill GBM cells via three manners.

SUMMARY:
The goal of this clinical trial is to learn if NRG103 works to treat recurrent GBM in adults. It will also learn about the safety of NRG103.

The main questions it aims to answer are:

Does NRG103 prolong overall survival or disease-free survival in patients with GBM? What medical problems do participants have when receiving NRG103 treatment? Researchers will give patients with NRG103 to see if NRG103 works to treat recurrent GBM.

Participants will:

Receive NRG103 twice in 14 days Visit the clinic once every 2 weeks for checkups and tests Keep a diary of their symptoms

DETAILED DESCRIPTION:
The annual incidence rate of malignant brain tumors in China is 4.2/100000, and GBM accounts for 50.9%. GBM is highly invasive and malignant. After undergoing anti-tumor treatments such as surgery, radiotherapy, and chemotherapy, the short-term recurrence rate is extremely high. The median survival time after recurrence is only 9 months, and the 1-year survival rate is 30%. It is urgent to explore new therapy strategy.

Transgenic oncolytic virus therapy for GBM is an emerging anti-tumor therapy. The genetically engineered oncolytic virus has improved selectivity towards tumor cells, replicating and lysing only within infected tumor cells, while activating the body's immune system to launch a more extensive attack on tumors. At present, various genetically modified oncolytic viruses targeting GBM have entered the clinical trial stage both domestically and internationally. For example, G47Δ, with superior anti-tumor activity and good safety in early clinical trials, has been conditionally approved for marketing in Japan for the treatment of malignant gliomas. DNX-2401, JL15003, and others are also in the early stages of clinical research. NRG-103 is an innovative gene therapy drug developed based on the in situ trans-differentiation technology. Through multiple mutation modifications of the adenovirus genome, it can enhance the specific recognition and killing effect of oncolytic virus on GBM tumor cells without being limited by tumor gene phenotype, and regulate the immune microenvironment to induce stronger anti-tumor immune response. In addition, the two transcription factors expressed on NRG-103 can efficiently transdifferentiate residual GBM tumor cells into non tumor like neuronal cells, in order to achieve the goal of delaying tumor recurrence and long-term survival. NRG-103 exhibits significant anti-tumor activity and clear in situ trans-differentiation effects in preclinical models, providing scientific evidence for the potential clinical efficacy of NRG-103.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years.
2. Patients must have histologically or cytologically confirmed glioblastoma(WHO 2021).
3. Patients have experienced recurrence (RANO 2.0) after previous anti-tumor treatments, including the recurrent tumor has been surgically removed and an Ommaya reservoir has been placed inside the tumor cavity.
4. The relevant adverse reactions from the previous treatment have been restored to ≤1 level(NCI-CTCAE v5.0).
5. Karnofsky Performance Score≥70.
6. Stable doses of dexamethasone during the week prior to inclusion.
7. Adequate bone marrow reserve: White blood cell count>2.0 × 109/L, neutrophil count>1.0 × 109/L, platelet count>100 × 109/L, international normalized ratio ≤1.5 times ULN, and activated partial thromboplastin time≤1.5 times ULN.
8. Normal heart, renal and liver function.
9. Effective method of contraception for patients and their partners.
10. Written informed consent.

Exclusion Criteria:

1. Allergy to the components of the test drug and contrast agent.
2. Unable to undergo imaging examinations required for the research.
3. A history of cell therapy, gene therapy, or oncolytic virus therapy.
4. Undergoing other clinical trials.
5. A history of anti-tumor vaccines or other immunomodulatory drugs with 4 weeks.
6. A history of other type of malignant tumors.
7. Unexplained fever.
8. A history of autoimmune disease.
9. A history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
10. Active hepatitis B, or hepatitis C.
11. Severe heart disease (NYHA III or IV), or poorly controlled diabetes.
12. Two or more GBM lesions.
13. GBM lesion located in the brainstem, cerebellum, posterior fossa, or spinal cord, as well as leptomeningeal diseases.
14. A history of diffuse subarachnoid and subarachnoid diseases.
15. GBM lesion invades the ventricular wall or tumor cavity communicates with the ventricle after surgery.
16. A history of encephalitis, multiple sclerosis, or other central nervous system infections.
17. Cerebral herniation syndrome.
18. Pregnant and lactating women.
19. Other situations that the researcher deems unsuitable for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months after NRG-103 treatment
  The participants will be followed until disease progression by RANO criteria

SECONDARY OUTCOMES:
Overall survival | 12 months after NRG-103 treatment
  The participants will be followed until death

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Li, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Data related to this clinical trial will be protected by Zhongnan Hospital